CLINICAL TRIAL: NCT03525054
Title: Semantic and Syntactic Computerized Analysis of Free Speech
Acronym: ASESID
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ASESID (29BRC17.0198)
Record Dates: First submitted 2018-04-26; First posted 2018-05-15 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Psychotic Disorders; Psychosis; Schizophrenia and Related Disorders; Schizophrenia Prodromal; Diagnosis, Psychiatric
Keywords: Psychotic Disorders; Diagnosis, Psychiatric; Schizophrenia Prodromal; Ultra High Risk; Prediction Of Psychosis; Machine Learning; Automated Language Analysis; Semantic Coherence; Syntaxic Complexity
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Schizotypal Personality Disorder; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Subtle speech disorganization could be predictive of a transition to schizophrenia of ultra-high-risk patients. The aim of our longitudinal multicenter cohort study is to identify specific linguistic markers of the psychotic transition to validate a french predictive model of this transition using computerized speech analysis techniques

DETAILED DESCRIPTION:
Different scales allow identification of patients at ultra-high-risk to develop psychosis. The current challenge is to identify a predictive marker of transition to schizophrenia. Language disorders, which reflect psyche, could be one of these markers. Computerized speech analysis techniques such as Latent Semantic Analysis (LSA) have already proven their reliability in schizophrenia. These techniques reveal subtle speech disorganization that would be predictive of a clinical transition of ultra-high-risk psychotic patients. A combination of semantic and syntactic analysis could accurately predict the psychotic transition. The aim of our longitudinal multicenter cohort study is to validate this predicitve model in french language as well as identifying specific linguistic markers of the psychotic transition.

The initial report including the CAARMS is completed with an audio recording from the initial medical interview. The recording will be transcribed and analyzed by computer following the method of lemmatization and vectorial analysis (LSA). An analysis of the grammatical function (number of words, rate of the various grammatical functions) will also be performed. This first analysis will emerge linguistic markers correlated to transition to psychosis that we will use to construct a predictive model for transition to schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Major and/or minor from 15 to 30 years old
* Who alleged a suicidal gesture or idea or behavior that has repercussions in their emotional, social or professional life
* If patients receive neuroleptic treatment that impairs cognitive abilities, a one-week wash-out period will be scheduled prior to assessment.

Exclusion Criteria:

* History of psychosis
* Risk of self-harm or violence not compatible with outpatient treatment
* QI<70 (WAIS)
* Neurological disorder or major health problem
* Impossibility to interrupt neuroleptic treatment for one week
* Refusal to participate

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Help-seekers patients are recruited during two years from the early psychosis detection centers in Brest, France (CEVUP), Paris, France (CJAAD) and in Lausanne, Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2028-05-02 (Estimated); Study Completion 2028-05-02 (Estimated)

PRIMARY OUTCOMES:
Transition to schizophrenia | 2 years
  Determined from the CAARMS scale (COMPREHENSIVE ASSESSMENT OF AT RISK MENTAL STATES)

SECONDARY OUTCOMES:
Identification of patients at "ultra high risk " for developing schizophrenia | Day 0
  Determined from the CAARMS scale ( COMPREHENSIVE ASSESSMENT OF AT RISK MENTAL STATES)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHRU de Brest, Brest
  - Meunier Sophie, Caen
  - CH de SAINT ANNE, Paris

IPD SHARING:
Plan to Share IPD: No